CLINICAL TRIAL: NCT01109043
Title: b. p. m Study (Beats Per Minute): Heart Rate Development Whilst Treating Patients With Hypertension With Concor or Concor Plus
Brief Title: Bisoprolol in Hypertension: Effect on Concomitant Elevated Heart Rate
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Gesellschaft mbH, Austria (Industry)
Responsible Party: Sponsor
Other Study IDs: 084000-504
Record Dates: First submitted 2010-04-19; First posted 2010-04-22 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: Hypertension; Bisoprolol; Antihypertensive drugs; Blood pressure; Quality of life; Diabetes; Ketohexokinase
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Bisoprolol; Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Bisoprolol or bisoprolol + HCTZ — Film-coated tablets containing 5 mg or 10 mg of bisoprolol hemifumarate or film-coated tablets containing 5 mg of bisoprolol fumarate (2:1) and 12.5 mg of HCTZ were given
  Other Names: Concor or Concor Plus

SUMMARY:
The b.p.m study will be performed to gain the insight in the courses of illness and therapy in subjects, suffering from hypertension and that have elevated heart rate. This study will show that a therapy with bisoprolol (Concor/Concor PLUS) or any other blood pressure lowering (antihypertensive) drug lowers blood pressure (BP) and heart rate and increases the quality of subjects' life.

DETAILED DESCRIPTION:
The b.p.m study measures heart rate development whilst treating subjects with hypertension with Concor [bisoprolol] or Concor Plus [bisoprolol + hydrochlorothiazide (HCTZ)].

The objectives of this study are:

After 6 months of the therapy treatment, 60% of the subjects showed a heart rate ≥ 80 beats/min.

An improved quality of life information after 6 months of therapy treatment, collected by asking standardised questions A decrease in systolic and diastolic BP after 6 months presented significant differences Digital sphygmomanometers (BP measuring devices) will be supplied in order to document the values of BP and heart rate. Blood pressure and heart rate should be measured at least 2 times, ideally 4 times per day. Furthermore, every subject will additionally receive a documentation sheet, where he/she will record the measurement data. The documentation sheet will be a part of the improvement of the quality of life; it can be removed and passed on.

Every subject will be explained how to use and handle the BP measuring device and the importance of the documentation. The assessment of the quality of life must be made at the beginning and at the end of 6 month therapy. Within the framework of the examination the attending physician will ask 8 standard questions (SQ-8 Short Form Health Survey). The questionnaire will be a part of the quality of life assessment.

The main focus of the observation is on the age group < 55 years with concomitant diseases, such as diabetes or ketohexokinase (KHK).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with high blood pressure (BP) and tachycardia
* Subjects with essential hypotonia, angina pectoris
* Subjects with essential hypertonia, when a therapy with ß-blockers or diuretics is not sufficiently effective
* Precautions to be taken in case of severe peripheral circulation disorders, diabetes (especially at the time, when blood sugar is elevated), during a strict fast, in case of metabolic acidosis, atrioventricular block (AV) block of grade I, Prinzmetal angina, additional therapy with angiotensin-converting enzyme inhibitors (ACE-inhibitors), severe coronary or cerebral sclerosis, hyperuricemia or gout and in subjects with a history of severe hypersensitive reactions or during a desensitization therapy (excessive anaphylactic reaction, attenuated adrenergic counterregulation)
* Special precautions must be taken with the subjects that have a family history or suffered from psoriasis, during a desensitization therapy (also anamnestic subjects), other obstructive pulmonary diseases on account of the possibility of initiation or intensification of bronchoconstriction, although, due to the marked ß1-selectivity of bisoprolol, the risk is lower than with non-selective ß-receptor blockers. The subjects that have a family history or suffered from psoriasis should the take Concor Plus only after a careful assessment of risk - benefit ratio. The subjects with pheochromocytoma should take Concor Plus, as well as other ß-blockers after inhibiting the alpha-receptors

Exclusion Criteria:

* Subjects with acute cardiac insufficiency, sinus sick syndrome, bradycardia and anaemia
* Contraindicated medical conditions for bisoprolol as defined in the Product Information, i.e. a known hypersensitivity to the active agent bisoprolol or one of the inactive ingredients of the medication; acute heart failure or decompensation of heart insufficiency, that requires a therapy with inotropic agents; cardiogenic shock; AV block grade II or III (in the absence of cardiac pacemakers); sick sinus syndrome, sinoatrial heart block; symptomatic bradycardia; symptomatic hypotonia; severe asthma bronchiolus or severe chronic obstructive airways disease; advanced stages of peripheral arterial disease or Raynaud's Syndrome; untreated pheochromocytoma, metabolic acidosis
* Contraindicated medical conditions for bisoprolol + hydrochlorothiazide (HCTZ) as defined in the Product Information, i.e. hypersensitivity to the ingredients of the medication containing bisoprolol + HCTZ, uncompensated heart insufficiency, pulmonary hypertension, cardiogenic shock, AV block, grades II and III. sick sinus syndrome (in the absence of cardiac pacemakers), sinoatrial heart block, severe bradycardia with less than 50 beats/min from the start of treatment, hypotension(systolic less than 90 mmHg), acute asthmatic attack, intravenous administration of calcium antagonists of Verapamil type, simultaneous treatment with monoamine oxidase inhibitors (MAO-inhibitors), advanced stages of peripheral circulation disorder, severe therapy-resistant potassium deficiency, severe hyponatraemia, hypercalcaemia, severe renal dysfunction (serum creatinin over 1.8 mg/100 ml and/or creatinin clearance under 30 ml/min); acute glomerulonephritis; liver coma; children, not previously treated; pregnancy and breastfeeding

Max Age: 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Hypertensive subjects
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Improvement in heart rate | Baseline to 6 months of therapy treatment
Changes in systolic and diastolic BP | Baseline to 6 months of therapy treatment

SECONDARY OUTCOMES:
Assessment of quality of life (SQ-8 Short Form Health Survey) | Beginning and at the end of 6 month therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard List, Study Director — Merck Serono Austria a division of Merck Gesellschaft mbH, Austria, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Merck Serono Research Site, Vienna, Austria